CLINICAL TRIAL: NCT05751304
Title: A Comparative Study Between Intrathecal Dexmedetomidine VS Ketamine With Intrathecal Bupivacaine in Orthopedic Lower Limb Surgeries.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ziad Ahmed Ali, A comparative study between intrathecal dexmedetomidine VS ketamine with intrathecal bupivacaine in orthopedic lower limb surgeries., Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-02-09
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Bone Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Active Comparator): (50 patients) will receive calculated dose of intrathecal hyperbaric bupivacaine 0.5 % according to body weight and 5μg dexametomidine.
  Interventions: Drug: Dexmedetomidine
- Group K (Active Comparator): (50 patients) will receive calculated dose of intrathecal hyperbaric bupivacaine 0.5 % according to body weight and 0.1 mg/kg ketamine.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — (50 patients) will receive calculated dose of intrathecal hyperbaric bupivacaine 0.5 % according to body weight and 5μg Dexametomidine.
  Arms: Group D
Drug: Ketamine — (50 patients) will receive calculated dose of intrathecal hyperbaric bupivacaine 0.5 % according to body weight and 0.1 mg/kg ketamine.
  Arms: Group K

SUMMARY:
Orthopedic anaesthesia and acute postoperative pain management, two anesthesiology subspecialties,are getting more credit for reducing hospital stays, promoting functional recovery and improving patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

-The study will include 100 adult patients (18 to 50 years old) with ASA physical status class I and class II undergoing orthopedic lower limb surgeries under itrathecal anathesia .

Exclusion Criteria:

* Patient refusal.
* Drug abuse.
* Patient with neurological, psychiatric or neuromuscular disease.
* Chronic pain on medicine.
* Known allergy to the study medications.
* Patients e contraindications to intrathecal anesthesia .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
comparison between duration of analgesia from Ketamine Vs Dexmedtomidine in the Patients with lower limb surgery | 1 year
  comparison between duration of analgesia from Ketamine Vs Dexmedtomidine in the Patients with lower limb surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Kehlet H, Holte K. Effect of postoperative analgesia on surgical outcome. Br J Anaesth. 2001 Jul;87(1):62-72. doi: 10.1093/bja/87.1.62. No abstract available. PMID 11460814
- [Background] Brennan F, Carr DB, Cousins M. Pain management: a fundamental human right. Anesth Analg. 2007 Jul;105(1):205-21. doi: 10.1213/01.ane.0000268145.52345.55. PMID 17578977